CLINICAL TRIAL: NCT06257602
Title: Tragal Cartilage Graft Tympanoplasty: Microscopic Versus Endoscopic
Brief Title: Microscopic Versus Endoscopic Tympanoplasty
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rania Tharwat Fahmi, Director, Assiut University
Other Study IDs: Endoscopic tympanoplasty
Record Dates: First submitted 2023-12-07; First posted 2024-02-14 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic tympanoplasty group: Endoscopc tympanoplasty group: rigid endoscope 3 mm diameter/14 cm long/0 angle of view will be used together with a high-definition camera head and monitor and using tragal graft to reconstruct perforations of tympanic membrane.
  Interventions: Procedure: Tragal graft tympanoplasty
- Microscopic tympanoplasty group: Microscopic tympanoplasty group: operating microscope and microscopic instruments will be used, and using tragal graft to reconstruct tympanic membrane perforations.
  Interventions: Procedure: Tragal graft tympanoplasty

INTERVENTIONS:
Procedure: Tragal graft tympanoplasty — Comparison study between Endoscopic and microscopic tympanoplasty using tragal graft
  Other Names: Endoscopic tympanoplasty

SUMMARY:
In this study, The investigatirs will compare surgical and anatomical outcomes of endoscopic and microscopic tympanoplasty type 1(myringoplasty) using tragal perichondrum and cartilage, and conduct a post-treatment survey regarding:

1. Graft uptake, hearing outcome, postoperative pain, and healing time.
2. Assess the operation time.

DETAILED DESCRIPTION:
Tympanic membrane perforation repair or tympanoplasty is a successful technique and has been validated in numerous studies since Wullstein and Zollner first proposed it in 1952. Previously, the technique was performed with illumination and magnification under a microscope. It typically requires an extensive postauricular incision to get through the narrow and curved external auditory canal, especially in child, complex perforations. The exclusive transcanal endoscopic tympanoplasty technique emerged in the 1990s; it provides more direct and wider surgical viewing angle, and it largely reduces the necessity for a traumatic postauricular incision in difficult cases. It has been gaining ground rapidly in recent years. Although closure rates tympanoplasty surgery can reach 90% or more, higher failure rates are seen in children, larger perforations, chronic Eustachian tube dysfunction, and in bilateral cases. Postoperative improvement in hearing is closely related to the postoperative change in the tympanogram. Postoperative hearing results and tympanograms are mainly influenced by the mucosal condition of the Eustachian tube (ET) orifice. Relatively greater improvement in hearing is observed in the long-term follow- up. Different graft materials have been proposed over the years to improve surgical outcomes, the search for an ideal graft is a subject of continued discussion, as transcanal endoscopic approaches have been proposed for larger and more complex perforations once reserved for postauricular techniques. The temporalis fascia (TF) has been the most preferred graft material for conventional microscopic tympanoplasty via postauricular or endaural approaches; it has theadvantages of having a readily available and plentiful source, and though its durability has been challenged in recent years, it is still widely used. However, with the increasing popularity of transcanal endoscopic ear surgery (TEES), an increasing number of otologists have adopted this technique and switched to using the nearby tragal perichondrium/cartilage graft when the surgical route is changed. The tragus has a pivotal function in reconstruction in ear surgery, and it is limited in source; hence, harvest on an ad hoc basis may lead to donor insufficiency at ensuing surgeries. Moreover, the tragus constitutes the anterior cartilaginous skeleton of the EAM and plays a role in sound transmission; maintaining its integrity would benefit future hearing device applications.

ELIGIBILITY:
Inclusion Criteria:

* Inactive chronic tubotympanic otitis media (dry ear: no otorrhea without

medication for at least 1 month).

* Patients with age 15-45 years old in both sexes.
* Patients with pure conductive hearing loss. unhealed tympanic membrane perforation for >3 months.
* Patients who are willing to give consent for the study.

Exclusion Criteria:

* Deeper lesions (Attico-antral disease, ossiculopathy, atelectasis, cholesteatoma, etc.), if suspected, on computed tomography scan.
* Patients below 15 years old, and more than 45 years old.
* Previous tympanoplasty, or other ear surgery.
* Sensori- neural hearing loss.
* Discharging ear.
* Narrow obvious narrowing of the EAC or syndromes that affect the middle ear (e.g., Down syndrome). 7) Comorbid systemic diseases like diabetes or any chronic specific infection.

Ages: 15 Years to 45 Years | Sex: All
Age Groups: Child, Adult
Study Population: After fulfilling all inclusion and exclusion criteria all patients will be subjected to
  * Full history taking including:
  * Personal History.
  * Full medical history includes: onset, course, duration, last attack, amount, and color of otorrhea.
  * History of hearing loss, tinnitus, and vertigo.
  * History of previous ear surgery.
  * Nasal symptoms, and other otorhinology symptoms.
  * Full otorhinology examination:
  * Full otorhinology examination including:
    1. Otological assessment: Size, site, side of perforation, and any ear discharge or any abnormality of the external auditory canal.
    2. Hearing tests.
    3. Nasal examination.
  * Audiological evaluation: (before and after surgery):
  * Pure tone audiometry.
  * Impedance tympanogram.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Tragal cartilage graft tympanoplasty: Microscopic versus endoscopic | 24 months
  Time taken during surgery in microscopic tympanoplasty versus time taken during endoscopic tympanoplasty in minutes

REFERENCES:
- [Background] Thomassin JM, Duchon-Doris JM, Emram B, Rud C, Conciatori J, Vilcoq P. [Endoscopic ear surgery. Initial evaluation]. Ann Otolaryngol Chir Cervicofac. 1990;107(8):564-70. French. PMID 2085261